CLINICAL TRIAL: NCT03583281
Title: Effects of Dietary Fatty Acids on Octadecanoid Production and Biological Actions in Obesity-induced Inflammation: Implications for Dietary Requirements
Brief Title: Effects of Dietary Fatty Acids on Octadecanoid Production and Biological Actions in Obesity-induced Inflammation
Acronym: OXBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H18926
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Intervention Model Description: Obese females
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flax oil (Active Comparator): Participants will consume capsules containing flax oil (4 grams alpha-linolenic acid [ALA] per day) for 4 weeks
  Interventions: Dietary Supplement: Capsules containing flax oil
- Fish oil (Active Comparator): Participants will consume capsules containing DHA-enriched fish oil (4 grams DHA per day + 0.8 grams EPA per day) for 4 weeks
  Interventions: Dietary Supplement: Capsules containing DHA-enriched fish oil

INTERVENTIONS:
Dietary Supplement: Capsules containing flax oil — Capsules containing flax oil to provide 4 grams ALA per day for 4 weeks
  Arms: Flax oil
Dietary Supplement: Capsules containing DHA-enriched fish oil — Capsules containing fish oil to provide 4 grams DHA per day and 0.8 grams EPA per day for 4 weeks
  Arms: Fish oil

SUMMARY:
This is a single site, double-blind, randomized, crossover study designed to compare the effects of dietary supplementation with flax oil rich in alpha-linolenic acid (ALA) and fish oil rich in docosahexaenoic acid (DHA) on oxylipin profiles over time (0 to 4 weeks) and among obese females varying in their inflammatory state. Additional assessments will include plasma fatty acid composition, adipokines, markers of adipocyte dysfunction and inflammation; immune cell/monocyte fatty acid composition, and functional properties including their metabolism and oxylipin production; and vascular function.

DETAILED DESCRIPTION:
A single site, double-blind, randomized, cross-over study designed to compare the effects of flax oil and fish oil supplementation on the oxylipin profile in females with obesity (n=24). Eligible participants will complete two supplementation phases (flax oil and fish oil rich in DHA) and will be asked to attend 3 in-person clinic visits (0, 3, and 28 days) for blood and urine collection during each phase. In addition to oxylipin profiles, assessments will include plasma fatty acid composition, adipokines, markers of adipocyte dysfunction and inflammation; immune cell/monocyte fatty acid composition, and functional properties including their metabolism and oxylipin production; and vascular function. If participants sign an optional consent form, vaginal fluid samples will be obtained at 0 and 28 days of each Supplementation Phase and analyzed for oxylipin and immune cell profile.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, non-lactating premenopausal female, >20 and <55 years of age (females of child bearing potential must take adequate birth control measures through the trial, and if a female becomes pregnant during the study, they must immediately stop taking the study oil capsules and be withdrawn from the study);
2. Fasting LDL-cholesterol ≤4.5 mmol/L and triglycerides ≤4.5 mmol/L (management with cholesterol-lowering and triglyceride-lowering medications is acceptable), plasma creatinine ≤265 µmol/L, AST <5× upper limit of normal (ULN) where the normal range is 10 - 32 U/L, ALT <5× ULN where the normal range is <25 U/L for females and <30 U/L for males, and glycated hemoglobin <6.5%;
3. Blood pressure <160/100 (management with anti-hypertensive medications is acceptable);
4. BMI ≥30, and waist circumference >94 cm for males and >80 cm for females of Asian ethnicity, and >102 cm for males and >88 cm for females of non-Asian ethnicity;
5. Stable regime if taking vitamin and mineral/dietary/herbal supplements for the past 1 month and while participating in the study;
6. Willing to maintain a stable level of activity while participating in the study;
7. Willing to maintain dietary routine and to refrain from consuming omega-3 supplements or omega-3 rich foods (>0.3 grams ALA/serving, or >0.1 grams EPA + DHA/serving), and to refrain from anti-inflammatory natural health products, from acceptance into the study until the final study visit;
8. Females must have normal menses and can be on birth control;
9. Agrees to not donate blood or blood products (e.g. platelets) while participating in the study and for 2 months after participation in the study;
10. Willing to comply with the protocol requirements and procedures;
11. Willing to provide informed consent.

Exclusion Criteria:

1. Has experienced a cardiovascular event (e.g. heart attack, stroke) or had a surgical procedure for cardiovascular disease (e.g. bypass, stent), presence of diabetes, chronic renal disease, liver disease (with exception of fatty liver), rheumatoid arthritis, immune disorder or disease (e.g. multiple sclerosis, leukemia), cancer in the previous 5 years, neurological disorders, gastrointestinal disorders or gastrointestinal surgery or bariatric surgery, or liposuction, or experiences migraines;
2. Taking medications for inflammation, pain or arthritis (e.g. cyclooxygenase (COX) inhibitors, steroids such as cortisone and prednisone), medications for blood glucose management, anti-coagulants/blood thinners, low dose acetylsalicylic acid, medication for erectile dysfunction (e.g. Viagra), within the last 3 months;
3. Regular use (> one day per week during two or more weeks) of acetylsalicylic acid (e.g. Aspirin), ibuprofen (e.g. Advil) or over-the-counter anti-inflammatory products such as Naproxen (e.g. Aleve, Midol Extended Relief) or those containing steroids such as cortisone and prednisone, within the last 3 months or while participating in the study;
4. Regular use (>three days per week during menstruation or >one day per week during two or more other weeks) of acetaminophen (e.g. Tylenol, Midol), within the last 3 months or while participating in the study;
5. Allergy or sensitivity to any of the study product ingredients, such as flax oil or flaxseed, fish oil or its sources such as fish or shellfish;
6. Cigarette/cigar smoking or use of tobacco products within the past 12 months or during the study;
7. Body weight has not been stable (plus or minus 3 kg) over the past 6 months;
8. Consumption of >15 alcoholic beverages per week (according to Canada's Low-Risk Alcohol Drinking Guidelines, 2012) within the last 3 months or while participating in the study;
9. Current (within the past 30 days) bacterial, viral or fungal infection;
10. Unable to obtain blood sample at the screening, week 0 visit, or two consecutive study visits;
11. Donated blood or blood products (e.g. platelets) or had blood collected in the 2 months prior to participation the study.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Plasma oxylipin concentrations over time | Baseline, 3 days, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0, 3 and 28 of each Supplementation Phase for the assessment of plasma oxylipin profile.

SECONDARY OUTCOMES:
Plasma fatty acid composition over time | Baseline, 3 days, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0, 3 and 28 of each Supplementation Phase for the assessment of plasma fatty acid composition.
Monocyte metabolism over time | Baseline, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0 and 28 of each Supplementation Phase Changes for isolation of monocytes and assessment of their metabolic characteristics evaluated by Seahorse.
Monocyte fatty acid composition over time | Baseline, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0 and 28 of each Supplementation Phase for isolation of monocytes and assessment of their fatty acid composition.
Peripheral blood mononuclear cell (PBMC) oxylipin and cytokine production over time | Baseline, 3 days, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0, 3, and 28 of each Supplementation Phase Changes for isolation of PBMCs and assessment of oxylipin and cytokine production ex vivo
Plasma adiponectin concentrations over time | Baseline, 3 days, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0, 3 and 28 of each Supplementation Phase for the assessment of plasma adiponectin, an anti-inflammatory adipokine and marker of adipocyte dysfunction.
Vascular function changes over time | Baseline, 28 days
  Assessment of of vascular function using pulse wave velocity determined at Day 0 and 28 of each Supplementation Phase.
Plasma lipid profile, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine over time | Baseline, 3 days, 28 days
  A fasting venous blood sample will be obtained from participants on Days 0, 3, and 28 of each Supplementation Phase for the assessment of plasma lipid profile, ALT, AST and creatinine
Vaginal fluid oxylipin profile over time | Baseline, 28 days
  If participants sign an optional consent form, vaginal fluid samples will be obtained at 0 and 28 days of each Supplementation Phase for assessment of the concentrations of oxylipins.
Vaginal fluid immune cell composition and function over time | Baseline, 28 days
  If participants sign an optional consent form, vaginal fluid samples will be obtained at 0 and 28 days of each Supplementation Phase for characterization of immune cells by cell type and by functional assays for susceptibility to infection ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Carla G Taylor, PhD, Principal Investigator — St Boniface Research Centre
Locations (1):
- I.H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pauls SD, Rodway LR, Sidhu KK, Winter T, Sidhu N, Aukema HM, Zahradka P, Taylor CG. Oils Rich in alpha-Linolenic Acid or Docosahexaenoic Acid Have Distinct Effects on Plasma Oxylipin and Adiponectin Concentrations and on Monocyte Bioenergetics in Women with Obesity. J Nutr. 2021 Oct 1;151(10):3053-3066. doi: 10.1093/jn/nxab235. PMID 34293124